CLINICAL TRIAL: NCT04604301
Title: Clinical Evaluation of High Strength Zirconia-Reinforced Lithium Silicate Chairside CAD/CAM Crowns
Brief Title: Celtra Quatro Crown Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Principal Investigator, Dennis J. Fasbinder, DDS, Clinical Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00155462
Record Dates: First submitted 2020-10-22; First posted 2020-10-27 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-01

CONDITIONS: Fractured Tooth; Decayed Tooth; Unsatisfactory Restoration of Tooth
Keywords: Crown; Ceramic; CAD/CAM
MeSH Terms: conditions — Tooth Fractures

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The final thickness of the restoration was not identified until before treatment started The final cement was not identified in the treatment process until the crown was milled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Crown, 1.0mm thickness, Calcium Aluminate Ionomer Cement (Experimental): occlusal thickness of 1.0 mm delivered with a conventional Calcium Aluminate Ionomer cement
  Interventions: Device: Celtra Quatro
- Crown, 1.5mm thickness, Calcium Aluminate Ionomer Cement (Experimental): occlusal thickness of 1.5 mm delivered with a conventional Calcium Aluminate Ionomer cement
  Interventions: Device: Celtra Quatro
- Crown, 1.0mm thickness, dual cure resin cement (Experimental): occlusal thickness of 1.0 mm delivered with Prime and Bond elect Universal Bond in total etch mode with a dual cure resin cement
  Interventions: Device: Celtra Quatro
- Crown, 1.5mm thickness, dual cure resin cement (Experimental): occlusal thickness of 1.5 mm delivered with Prime and Bond elect Universal Bond in total etch mode with a dual cure resin cement
  Interventions: Device: Celtra Quatro

INTERVENTIONS:
Device: Celtra Quatro — Full ceramic crowns will be made from the high strength ceramic, Celtra Quatro

SUMMARY:
This investigation will be a clinical trial to study the performance of a newly developed high strength ceramic material for crowns. The ceramic has been approved by the FDA for patient treatment. A computer technique will be used to fabricate the crowns in a single appointment without the need for a temporary crown or second appointment. Two adhesive resin cement techniques will be used to hold the crown to the tooth and they will be evaluated for creating sensitivity to the tooth. The purpose of the study is to measure how well the high strength crowns function over an extended period of time.

DETAILED DESCRIPTION:
A recently introduced high strength, zirconia-reinforced lithium silicate (ZLS) ceramic material for full contour CAD/CAM crowns is reported to offer a more translucent and esthetic high strength crown in a more efficient oven firing process. Celtra Quatro (Dentsply Sirona) is submitted to a high temperature matrix firing cycle in the SpeedFire oven (Dentsply Sirona) to achieve high strength in less than 5 minutes following milling. It has a reported flexural strength of 650 MPa compared to 450 MPa for lithium disilicate glass ceramic and > 900 MPa for 3mol% full contour zirconia.

Most glass ceramic materials have a recommended material thickness of 1.5 mm to maximize the strength potential of the material. Occlusal reduction resulting in a crown thickness of 1.0 mm, equitable to the recommendation for full contour zirconia crowns, may be considered sufficient to maintain the desired high strength attained by the ZLS material. This would also result in a more conservative tooth preparation.

Another potential advantage of high strength ZLS crowns to many clinicians is that they may be inherently strong enough to allow for conventional cementation. However, for less retentive preparations, it may also be possible to adhesively bond the crowns through the use of adhesive resin cements.

It is the intent of this investigation to evaluate the clinical application and performance of the new high strength, zirconia-reinforced lithium silicate material (Celtra Quatro) for CAD/CAM-generated chair-side crown applications. Patients will be recruited to have 60 Celtra Quatro crowns prepared and delivered during a single dental appointment using a chairside CAD/CAM system (CEREC/Dentsply Sirona). The crowns will be recalled at 6 months and then yearly for 5 years to evaluate long-term outcomes of the crowns.

ELIGIBILITY:
Inclusion Criteria:

* must have at least one carious lesion or defective restoration or fractured tooth in a molar or premolar
* reason for restoration should extend more than one-half the intercuspal width of the tooth requiring a full crown restoration
* Teeth to be vital and asymptomatic prior to treatment
* No more than two restorations will be placed per patient. If a patient presents with more than two acceptable teeth for the study, molar teeth will be included prior to premolar teeth.

Exclusion Criteria:

* Devital or sensitive teeth
* Teeth with prior endodontic treatment of any kind
* Teeth with a history of direct or indirect pulp capping procedures
* Patients with significant untreated dental disease to include periodontitis and rampant caries
* Pregnant or lactating women
* Patients with a history of allergies to any of the materials to be used in the study
* Patients unable to return for the recall appointments

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Crown failure | from delivery of the crown up to 5 years
  Restoration failure is scored by visual loss of the crown from the tooth requiring replacement of the study crown with a new crown at any time between delivery and five years.

SECONDARY OUTCOMES:
Crown loss of retention | from delivery of crown up to 5 years
  Loss of retention is measured as visual detachment or dislodgment of the crown from the tooth without fracture of the crown requiring recementation of the crown at any time between delivery and five years.
Tooth sensitivity | from delivery of crown up to 5 years
  Patient described sensitivity on a scale of 1 to 4, where 1 means absence of sensitivity (pain) and four means severe discomfort noted routinely with cold or pressure stimulation.
Margin staining | from delivery of crown up to 5 years
  Margin staining is categorized based on modified US Public Health Service criteria using a four point scale where 1 is no staining and 4 is penetrating stain involving more than 50% of the margin.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Fasbinder, DDS, Principal Investigator — University of Michigan
Locations (1):
- School os Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No